CLINICAL TRIAL: NCT05857293
Title: Outcomes for Patent Ductus Arteriosus Stenting in Neonates With Duct-Dependent Pulmonary Circulation: A Prospective Study at Sohag University Hospital
Brief Title: PDA Stent in Neonates With PDA Dependent Pulmonary Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Somia Sabry Mahmoud, Assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-04-03MD
Record Dates: First submitted 2023-05-02; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Neonatal Cyanosis Due to PDA Dependent Pulmonary Circulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyanotic neonate (Experimental): Cyanotic neonates with PDA dependent pulmonary circulation will be treated with catheter guided PDA stent implantation to keep duct patency and improve oxygen saturation
  Interventions: Device: Catheter-guided PDA stent implantation

INTERVENTIONS:
Device: Catheter-guided PDA stent implantation — PDA stent is the primary treatment for patients with duct-dependent pulmonary circulation. It serves as a temporary bridge for later surgical repair by keeping the duct patent to improve oxygen saturation
  Other Names: PDA stent

SUMMARY:
After echocardiography confirmation of PDA dependent pulmonary circulation in cyanotic neonates, catheter-guided PDA stent implantation will be done. Under general Anasthesia and after discontinuation of prostaglandin 4-6 hours before procedure, obtain vascular access and unfractionated heparin is given, then duct is accessed via a cut pig-tail or Judkins right [JR] catheter, and is crossed by PTCA wire to be carefully placed in the left or right branch pulmonary arteries, choose proper stent diameter and length, place the stent and confirm it's position, NICU admission for the neonate with heparin infusion for 24-48 hrs and acetylsalicylic acid is given then follow up the patient by pulse oximeter and echocardiography

ELIGIBILITY:
Inclusion Criteria:

Neonates and young infants with duct dependent pulmonary circulation

Exclusion Criteria:

* Untreated sepsis.
* Coagulopathy.
* PDA dependent systemic circulation.

Ages: 1 Hour to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oxygen saturation | Change in oxygen saturation within 24 hours
  Using pulse oximeter to assess oxygen saturation
Evaluation of duct patency | 1 month
  Using echocardiography assess flow through the duct

CONTACTS AND LOCATIONS:
Overall Officials: Somaia S Mahmoud, Master, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt